CLINICAL TRIAL: NCT00145444
Title: A Multicenter, Double-Blind, Randomized Trial Of Ziprasidone (80 - 160 Mg) Versus Olanzapine (10 - 20 Mg) In Patients With Recent-Onset Schizophrenia, Schizoaffective And Schizophreniform Disorder.
Brief Title: Kahn Study; Investigation Of The Efficacy Of Ziprasidone Versus Olanzapine In The Management Of Recent-Onset Psychosis; A Flexible-Dose, Parallel Group, Double-Blind Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1281006
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia; Psychotic Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine; ziprasidone

INTERVENTIONS:
Drug: olanzapine
Drug: ziprasidone

SUMMARY:
This study intends to compare novel antipsychotics ziprasidone and olanzapine, to confirm the findings of an open study -where stable patients receiving olanzapine switched to ziprasidone- which showed maintenance of clinical effect with improvements in all domains of cognitive function at 6 weeks (Daniel, 1999). Direct comparison of the two agents in a well-controlled double-blind fashion will allow an evaluation of the effect on cognitive function in the short and long-term management of patients with recent-onset schizophrenia, schizoaffective and schizophreniform disorder.

ELIGIBILITY:
Inclusion Criteria:

* Duration of illness < 5 years (according to DSM-IV and onset first psychotic episode); CGI severity score > 4 (moderately ill)
* maximum exposure to antipsychotic treatment of =< 16 weeks.

Exclusion Criteria:

* Concurrent treatment with antipsychotic agents =< 12 hours prior to randomization
* for depot agents a period of two weeks or one cycle, whichever is the longer, must occur between last administration and randomization
* Treatment with antidepressants or mood stabilizers =< 7 days of randomization
* for MAOIs and moclobemide this period must =< 2 weeks
* for fluoxetine =< 5 weeks

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100
Dates: Start 2003-03; Study Completion 2005-11

PRIMARY OUTCOMES:
The effect on cognitive function of ziprasidone and olanzapine in the management of recent-onset psychosis, measured as the difference in efficacy in a 8 week period from the baseline visit to the end of week 8 visit.

SECONDARY OUTCOMES:
- to demonstrate effect on cognitive function of ziprasidone and olanzapine in the management of recent-onset psychosis, measured as the difference in efficacy over a 24-week and one year period from baseline visit to the end of week 24 and week 52 visit

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Belgium (3):
  - Pfizer Investigational Site, Antwerp
  - Pfizer Investigational Site, Duffel
  - Pfizer Investigational Site, Kortenberg
- Netherlands (4):
  - Pfizer Investigational Site, Ermelo
  - Pfizer Investigational Site, Groningen
  - Pfizer Investigational Site, Nijmegen
  - Pfizer Investigational Site, Utrecht

REFERENCES:
- [Derived] Grootens KP, van Veelen NM, Peuskens J, Sabbe BG, Thys E, Buitelaar JK, Verkes RJ, Kahn RS. Ziprasidone vs olanzapine in recent-onset schizophrenia and schizoaffective disorder: results of an 8-week double-blind randomized controlled trial. Schizophr Bull. 2011 Mar;37(2):352-61. doi: 10.1093/schbul/sbp037. Epub 2009 Jun 19. PMID 19542525
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281006&StudyName=Kahn+Study